CLINICAL TRIAL: NCT01654172
Title: Effect of Flavanol-rich Cocoa on Peripheral and Cerebral Blood Flow in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 05/Q2401/146
Record Dates: First submitted 2012-07-25; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes
Keywords: Diabetes; peripheral neuropathy; Cocoa flavanols
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Flavanol Cocoa (Experimental): Cocoa drink containing ~450mg cocoa flavanols and 10g carbohydrate per serving.
  Subject consumes 2 servings per day, for 7 days.
  Interventions: Dietary Supplement: High Flavanol Cocoa
- Low Flavanol Cocoa (Placebo Comparator): Cocoa drink containing ~25mg cocoa flavanols and 10g carbohydrate per serving.
  Subject consumes 2 servings per day, for 7 days.
  Interventions: Dietary Supplement: Low Flavanol Cocoa

INTERVENTIONS:
Dietary Supplement: High Flavanol Cocoa — Total daily flavanol intake provided by the high flavanol drink is ~900mg
  Arms: High Flavanol Cocoa
Dietary Supplement: Low Flavanol Cocoa
  Arms: Low Flavanol Cocoa

SUMMARY:
Cocoa flavanols form part of the family of chemicals (also found in red wine and tea) which have aroused interest due to population studies suggesting that diets high in these substances might reduce risks of heart disease. In the laboratory, these flavanols have been shown to cause blood vessels to widen and blood flow to increase. As dysfunction in this ability of blood vessels to widen is now thought to play a central role in the complications of diabetes, novel ways to mitigate this are constantly being sought.

The present study aims to use non-invasive magnetic resonance imaging (MRI) to measure foot and brain blood flow before and after 7 days consumption of a cocoa drink high in flavanols, in subjects with diabetes, with and without peripheral neuropathy.

DETAILED DESCRIPTION:
Cocoa flavanols form part of the family of polyphenols (also found in red wine and tea) which have aroused interest due to epidemiological studies suggesting that diets high in these substances might reduce risks of heart disease. However, it is difficult to account for all sources of polyphenols in these epidemiological studies, and the level of cocoa product consumption was generally not well documented. Furthermore, in readily available cocoa products, processing may remove most of the flavanols, leading to such products varying considerably in flavanol content. Recently, laboratory studies of the effects of cocoa flavanols have suggested an effect on the relaxation of smooth muscle in blood vessel walls, specifically the element mediated by the endothelium (blood vessel wall). Studies using ultrasound methods in healthy volunteers have shown an increase in blood flow in the arm following temporary arterial occlusion.

As endothelial dysfunction is now thought to play a central role in the complications of diabetes, novel ways to mitigate this are constantly being sought. It is well recognised that diabetic peripheral nerve damage leads to abnormal foot blood flow, including impaired superficial skin blood flow, and that this is one of the factors delaying wound healing in diabetic foot ulcers (the single largest cost in secondary care diabetes).

Several techniques are currently used to monitor blood flow to the limbs, including venous occlusion plethysmography (VOP), laser Doppler methods and nuclear medicine techniques. These techniques have low spatial resolution, low specificity, are labour intensive, or require the use of injected radioactive contrast agents (which pose a particular risk to diabetic patients). Radiation dose also limits repeat studies.

The arterial spin labelling magnetic resonance (ASL MR) technique is non-invasive, but yields a quantifiable measure of blood flow with high resolution, and allows measurements to be repeated several times, as the technique uses no external contrast agents.

The present study aims to use non-invasive magnetic resonance imaging (MRI) to measure peripheral (foot) and brain blood flow at baseline and in response to a cocoa drink high in flavanols, in subjects with type 2 diabetes, with and without peripheral neuropathy.

Subjects will attend an initial screening visit. Measures of HbA1c, kidney function and blood pressure will be checked, along with ankle-brachial pressure index (to check for poor circulation), foot pulses, and examination for peripheral nerve damage and cardiac neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Peripheral neuropathy or free from neuropathy

Exclusion Criteria:

* Current foot ulceration
* Hypertension
* Anti-hypertensive medications other than thiazide diuretics and ACE inhibitors
* Ischaemic heart disease
* Peripheral vascular disease (ABPI ,0.9 &/or impalpable foot pulses)
* Chronic kidney disease
* Poor glycaemic control
* DVT
* Epilepsy
* Pregnancy
* Contraindications to MRI
* Intolerance to lactose or cow's milk protein

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Brain Blood Flow | Day 0 and after 7d consumption of a cocoa drink
  Measured by ASL-MR at Day 0 and after 7d consumption of a cocoa drink to detect a change following intervention

SECONDARY OUTCOMES:
Change in Brain blood flow after acute consumption of cocoa | 1,3,5 and 8hrs after cocoa consumption
  Measured at day 0, (before intervention commences)and after 7days consumption of a cocoa drink
Change in Fasting foot blood flow | Day 0 and after 7d consumption of a cocoa drink
  Measured using ASL-MR
Change in Foot blood flow after acute consumption of cocoa | 1,3,5 and 8hrs after cocoa consumption
  Measured at day 0, (before intervention commences)and after 7days consumption of a cocoa drink
Change in Blood Flavanol concentration | Day 0 and after 7d consumption of a cocoa drink
  Measured at day 0, (before intervention commences)and after 7days consumption of a cocoa drink
Change in Fasting oxidative stress status | Day 0 and after 7 days of consuming a cocoa drink
  Oxidative stress assessed by measuring concentration of homocysteine, CRP, 8-isoprostaglandin, arginine and nitric oxide metabolites in the blood.
Change in diabetes control | Day 0 and after 7days of consuming a cocoa drink daily
  Assessment made from HbA1c, glucose and insulin concentration in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Simon Paige, MD, Principal Investigator — University Hospitals NHS Trust
Locations (1):
- University of Nottingham, Nottingham, Notts, United Kingdom